CLINICAL TRIAL: NCT01554917
Title: A Phase IV Study of Iguratimod in Patients With Active Rheumatoid Arthritis (RA)
Brief Title: A Study of Iguratimod in Patients With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIM-109
Record Dates: First submitted 2012-03-12; First posted 2012-03-15 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Iguratimod
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — iguratimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Iguratimod (Experimental)
  Interventions: Drug: Iguratimod

INTERVENTIONS:
Drug: Iguratimod — taken orally, 2 tablets/day (bid)

SUMMARY:
This study is intended to evaluate the safety and efficacy of Iguratimod in patients with active Rheumatoid Arthritis.

DETAILED DESCRIPTION:
This is a multi-center, open, single arm study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of RA
* Subjects who have active RA at the time of screening
* Subjects who haven't used any antirheumatic drugs or have used antirheumatic drugs for more than 3 months at the time of screening
* Written informed consent

Exclusion Criteria:

* Subjects with serious cardiovascular, renal, hematologic or endocrine diseases
* Pregnant or lactating women
* ALT>1.5×ULN, AST>1.5×ULN, Cr>135umol/L
* WBC<4×109/L，HGB<85g/L，PLT<100×109/L
* Subjects with uncontrolled infection
* Patients with active gastrointestinal diseases (such as gastric ulcer, etc.)
* Allergic to any of the study drugs
* History of alcoholism
* Subjects receiving live vaccines within 3 months prior to study entry
* Subjects participating in other clinical study within 3 months prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1759 (Actual)
Dates: Start 2012-05; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Percentage of patients meeting the American College of Rheumatology 20% response criteria (ACR20) | week 24
Incidence of adverse events | up to 28 weeks

SECONDARY OUTCOMES:
Percentage of patients meeting the American College of Rheumatology 50% response criteria (ACR50) | week 24
Percentage of patients meeting the American College of Rheumatology 70% response criteria (ACR70) | week 24
Change from baseline in Disease Activity Score 28 (DAS28) | week 24
Change from baseline in Health Assessment Questionnaire (HAQ) | week 24

CONTACTS AND LOCATIONS:
Overall Officials: Zhanguo Li, MD/PhD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mu R, Li C, Li X, Ke Y, Zhao L, Chen L, Wu R, Wu Z, Zuo X, Xie Y, Chen J, Wei W, Liu Y, Li Z, Dai L, Sun L, Liu X, Li Z. Effectiveness and safety of iguratimod treatment in patients with active rheumatoid arthritis in Chinese: A nationwide, prospective real-world study. Lancet Reg Health West Pac. 2021 Mar 22;10:100128. doi: 10.1016/j.lanwpc.2021.100128. eCollection 2021 May. PMID 34327344